CLINICAL TRIAL: NCT04203381
Title: Skeletal Health and Bone Marrow Composition Among Youth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amy DiVasta, MD (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor-Investigator, Amy DiVasta, MD, Chief, Division of Adolescent Medicine, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00033841
Record Dates: First submitted 2019-12-11; First posted 2019-12-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Gender Dysphoria in Children; Puberty; Bone Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transgender Participant (Other): Transgender children at Tanner stage II or early Tanner stage III between the ages of 9 and 14. Must be a current patient at a gender patient and within 6 weeks of initiating pubertal blockade treatment
  Interventions: Device: GnRH Agonist
- Cisgender Control Participant (No Intervention): Cisgender children Tanner II or early Tanner III between 9 and 14 matched by race, age, and BMI.

INTERVENTIONS:
Device: GnRH Agonist — Forty participants who are transgender and who have been prescribed a gonadotropin-releasing hormone (GnRH) agonist by their physician will undergo magnetic resonance imaging (MRI), magnetic resonance spectroscopy (MRS), dual-energy x-ray absorptiometry (DXA) and peripheral quantitative computed tomography (pQCT) scans at baseline, at 12 months and at 24 months after initiation of the GnRH agonist therapy. This longitudinal observational study of two cohorts seeks to identify significant changes in bone marrow adiposity and bone density over 24 months. The same assessments will be obtained in 40 healthy control subjects matched for age, race/ethnicity and body mass index, all factors that are known to influence skeletal outcomes. The evaluations of bone marrow adiposity will be correlated with bone density measurements and the assessments of mood (validated anxiety and depression scales) and health-related quality of life, before and after pubertal blockade.
  Other Names: Histrelin; Lupron; Pubertal Blockade
  Arms: Transgender Participant

SUMMARY:
Children and adolescents experiencing gender dysphoria feel increased distress with the onset of puberty. Gender clinics treat these young adolescents by "blocking" puberty using gonadotropin-releasing hormone (GnRH) agonist medications. This has the possibility of impacting bone development as sex steroids are important to bone mass development. In this multi-site study, the investigators will examine bone marrow composition (by MRI) in 40 transgender youth and bone density and body composition before/after pubertal blockade compared to healthy participants.

DETAILED DESCRIPTION:
The investigators propose to identify the effects of pubertal blockade on bone density and size in pediatric transgender individuals. Information is limited regarding bone health and metabolism for this group, and especially for children who are transgender. Further, the team's expertise in magnetic resonance imaging (MRI), magnetic resonance spectroscopy (MRS), dual-energy x-ray absorptiometry (DXA), and peripheral quantitative computed tomography (pQCT), examining the natal female skeleton in previous NIH funded studies, and extensive clinical expertise, provide an ideal foundation to apply this protocol to examine transgender female and transgender male skeleton. Findings from this study will allow us to identify potential preventative strategies to counter the long-term effects of puberty blockade such as osteoporosis and raise awareness of this medical consequence to medical care providers of transgender patients. The proposed project seeks to answer the clinically relevant question of how bone marrow composition relates to body composition, and its relation to both bone density and skeletal strength, in transgender patients who are undergoing puberty blockade, the first phase of therapy preceding gender-affirming hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing to give informed consent/assent (parent or legal guardian able to provide informed consent)
2. Tanner Stage II/III
3. Age 9-14 years old for assigned male at birth (AMAB) and 9-13 for assigned female at birth (AFAB)
4. Current patient at the Boston Children's Hospital Transgender Clinic or Cincinnati Children's Hospital Medical Center Clinic, within six weeks of initiating pubertal blockade treatment (e.g., GnRH agonist- Lupron or Vantas)
5. Controls are matched on age within 2 years, race/ethnicity, sex assigned at birth and BMI within 25%

Exclusion Criteria:

The participant must not:

1. Have chronic disease known to affect skeletal metabolism (e.g. cystic fibrosis, celiac disease, sickle cell disease, inflammatory bowel disease etc.)
2. Receipt of other medications within previous 3 months known to affect skeletal metabolism (e.g., glucocorticoids, anticonvulsants, etc.)
3. Have metal implants or hardware in their body that would not allow them to get an MRI
4. Have a diagnosis of a developmental disorder or claustrophobia that would prevent them from undergoing an MRI

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Participants must identify as transgender or nonbinary to be eligible for the study.
Enrollment: 80 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Bone marrow adiposity by magnetic resonance imaging (MRI) from baseline compared to 24 months | Change from baseline compared to 24 months
  Change from bone marrow adiposity measured by MRI (T1 maps) from baseline compared to 24 months
Change from magnetic resonance spectroscopy (MRS) from baseline compared to 24 months | Change from baseline compared to 24 months
  Change from T2 corrected fat/(fat+ water) ratios from baseline compared to 24 months

SECONDARY OUTCOMES:
Change from total body bone mineral density Z-score by Dual-energy X-ray absorptiometry (DXA) from baseline compared to 24 months | Change from baseline compared to 24 months
  Change from total body BMD Z-score from baseline compared to 24 months
Change from spine BMD Z-score by DXA from baseline compared to 24 months | Change from baseline compared to 24 months
  Change from lumbar spine BMD Z-score from baseline compared to 24 months
Change from hip BMD Z-score by DXA from baseline compared to 24 months | Change from baseline compared to 24 months
  Change from hip bone mineral density (g/cm2) from baseline compared to 24 months
Change from volumetric bone mineral density (vBMD) from baseline compared to 24 months | Change from baseline compared to 24 months
  Change from quantitative computed tomography (pQCT) scans will be obtained at sites 3%, 38%, and 66% of tibial length proximal to the distal growth plate from baseline compared to 24 months
Change from section modulus (bone bending strength) by quantitative computed tomography (pQCT) from baseline compared to 24 months | Change from baseline compared to 24 months
  Change from pQCT scans will be obtained at sites 3%, 38%, and 66% of tibial length proximal to the distal growth plate from baseline compared to 24 months

OTHER OUTCOMES:
Change from health-related quality of life (HRQL) from baseline compared to 24 months | Change from baseline compared to 24 months
  Change from HRQL will be assessed at initiation of the GnRH agonist, after 12 months and again after 24 months to understand the impact of pubertal blockade on quality of life using the validated survey, Child Health Questionnaire (CHQF)-87 from baseline compared to 24 months
Change from anxiety from baseline compared to 24 months | Change from baseline compared to 24 months
  Anxiety will be assessed at initiation of the GnRH agonist, after 12 months and again after 24 months to understand the impact of pubertal blockade on feelings of anxiety. Change from anxiety will be assessed using the validated survey, the SCARED from baseline compared to 24 months.
Change from depression from baseline compared to 24 months | Change from baseline compared to 24 months
  Change from depression will be assessed at initiation of the GnRH agonist, after 12 months and again after 24 months to understand the impact of pubertal blockade on feelings of depression using the validated survey, the Children's Depression Inventory (CDI-II) from baseline compared to 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No